CLINICAL TRIAL: NCT03345680
Title: Examining the Impact of School-based Dental Screening Program on Dental Visits and Dental Caries Among Primary School Children in Riyadh City, Saudi Arabia: A Randomized Controlled Trial
Brief Title: Examining the Impact of School-based Dental Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: King Saud University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: HR-16/17-4683
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2017-10

CONDITIONS: Dental Caries
Keywords: Dental visits; School-based program; Dental screening; Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Children will be screened, both parents and children will be informed of any abnormalities in the mouth.
- Interventional Group (Experimental): Interventional (Dental Screening) Children will be screened for dental caries and referred to a specific hospital for treatment, namely King Saud University Dental College, treatment will be provided free of charge to the referred participants.
  Interventions: Other: Referred to a specific hospital for treatment

INTERVENTIONS:
Other: Referred to a specific hospital for treatment — To King Saud University Dental College, treatment will be provided free of charge to the referred participants.
  Other Names: Interventional group
  Arms: Interventional Group

SUMMARY:
This study examines the effectiveness of school dental screening in promoting dental attendance and reducing untreated caries among primary schoolchildren in Riyadh, Saudi Arabia.

DETAILED DESCRIPTION:
Background: Dental caries is one of the most common diseases affecting children in Saudi Arabia despite the availability of free dental services. School-based dental screening could be a potential intervention that might impact uptake of service and subsequently dental caries.

Aim: To examine the effectiveness of school dental screening in promoting dental attendance and reducing untreated caries among primary schoolchildren in Riyadh, Saudi Arabia.

Methods: This is a cluster randomized controlled trial comparing referral of screened-positive children to a specific treatment facility (King Saud University Dental College Hospital) against the current practice (information letter advising parents to take their child to a dentist). A total of 1000 children in 12 schools will be recruited. Schools (clusters) will be randomly selected and allocated to either group using computer software. Clinical assessment for dental caries will be conducted at baseline and after 12 months by dentists using the World Health Organisation (WHO) criteria. Different clinical teams will be used for each trial group to ensure blinded outcome assessment. Data on socio-demographic, behavioural and dental visits will be collected at baseline and follow-up. Outcome measures will be the change in number of decayed teeth and the number of dental visits over 12 months.

Discussion: This project will use a robust design to provide high level of evidence on the clinical benefits of school dental screening. The findings will potentially inform policies related to the continuation/ implementation of school-based dental screening in Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 11 years (1st -5th grade at school) at baseline.
* Both Saudis and non-Saudis.
* Children for whom the person with parental responsibility has signed the consent form

Exclusion Criteria:

* Children in 6th grade (12-year-olds) as they would have left schools by the time of the follow-up assessment (12 months later).
* Children with any medically compromised condition such as congenital heart disease, haematological conditions, immune deficiency disease and end-stage renal disease.
* Children that refuse to participate (assent) in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 996 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
change in the number of decayed teeth (untreated caries) | 12 months
  the change in the number of decayed teeth (untreated caries) in both primary and permanent teeth 12 months after intervention.

SECONDARY OUTCOMES:
Changes in the proportion of children with untreated caries and whether the child visited the dentist | 12 months
  The change in the proportion of children with untreated caries in both deciduous and permanent teeth and whether the child visited the dentist

CONTACTS AND LOCATIONS:
Overall Officials: Haya M Alayadi, MSc, Principal Investigator — King's College London; Wael Sabbah, PhD, Study Director — King's College London
Locations (1):
- King's College London, London, Great Britin, United Kingdom

IPD SHARING:
Plan to Share IPD: No
data will not be shared except to central participant and principal investigator

REFERENCES:
- [Derived] Arora A, Kumbargere Nagraj S, Khattri S, Ismail NM, Eachempati P. School dental screening programmes for oral health. Cochrane Database Syst Rev. 2022 Jul 27;7(7):CD012595. doi: 10.1002/14651858.CD012595.pub4. PMID 35894680
- [Derived] Alayadi H, Sabbah W, Bernabe E. Effectiveness of school dental screening on dental visits and untreated caries among primary schoolchildren: study protocol for a cluster randomised controlled trial. Trials. 2018 Apr 13;19(1):224. doi: 10.1186/s13063-018-2619-2. PMID 29653545